CLINICAL TRIAL: NCT05277441
Title: A Novel Classification for the Assessment and Grading of Unexpected Events in Pediatric Surgery: The Clavien-Madadi Classification
Acronym: ComPedS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Omid Madadi-Sanjani, Dr., Principal investigator, Consultant Pediatric Surgery, Hannover Medical School
Other Study IDs: 9557_BO_K_2021
Record Dates: First submitted 2022-02-23; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Complication of Surgical Procedure; Complication of Anesthesia; Complication,Postoperative; Complication of Medical Care
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Novel severity grading system of unexpected events in pediatric surgery — Classification of unexpected events according to the Clavien-Madadi classification for pediatric surgical patients and simultaneously the non-modified Clavien-Dindo classification in more than 10.000 patients who have been treated at a single center from 2017 to 2022.

SUMMARY:
Postoperative adverse events may be associated with substantial morbidity and mortality. However, inconsistent definitions of complications and unexpected events have limited accurate analysis of surgical outcomes. In 2004, the Clavien-Dindo classification for postoperative complications has been introduced and has since then been validated in numerous studies, with more than 20.000 citations.

Despite the appraisal of the Clavien-Dindo classification in the pediatric surgical literature, some criticize the transfer of grading systems for adults into a pediatric cohort without modification or validation. In a recent study we have shown that few items of the classification do not offer relevant information in pediatric cohorts and we have added organizational and management errors, not integrated in the initial proposal by Dindo et al. Especially, the variety of options for the management of complications based on institutional protocols and logistics is emphasized and a more focused and detailed assessment of the invasiveness of procedures in children is introduced.

ELIGIBILITY:
Inclusion Criteria:

* All patients with unexpected events within the study period, treated at the department of pediatric surgery (preterms - 17 years of age), Hannover Medical School

Exclusion Criteria:

* None;

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Data on all patients (preterm infants to 18 years of age) who experienced unexpected events at the Department of Pediatric Surgery Hannover Medical School from 1st January 2017 to 31st December 2021 were documented prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through study completion, an average of 3 years

SECONDARY OUTCOMES:
Categorization of adverse events | Through study completion, an average of 3 years
  Events associated with surgical/non-surgical interventions and events not associated with interventions such as organizational problems, management problems or underlying disease were differentiated.
Classification of adverse events | Through study completion, an average of 3 years
  According to the Clavien-Dindo classification
Classification of adverse events using a novel instrument | Through study completion, an average of 3 years
  According to the Clavien-Madadi classification

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madadi-Sanjani O, Zoeller C, Kuebler JF, Hofmann AD, Dingemann J, Wiesner S, Brendel J, Ure BM. Severity grading of unexpected events in paediatric surgery: evaluation of five classification systems and the Comprehensive Complication Index (CCI(R)). BJS Open. 2021 Nov 9;5(6):zrab138. doi: 10.1093/bjsopen/zrab138. PMID 35022674